CLINICAL TRIAL: NCT00851539
Title: Educational Effectiveness of an HIV Pretest Video for Adolescents: A Randomized Controlled Trial
Brief Title: Evaluating Post-test HIV Counseling Videos for Teens
Acronym: Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Bronx Healthcare Network (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Yvette Calderon,MD, MS, Professor of Clinical Emergency Medicine, North Bronx Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2006-443; 5K23HD054315 (NIH)
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: HIV; HIV Infections
Keywords: HIV; Teenagers; Adolescent; HIV Testing; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Participants received counseling from a live counselor.
- Video (Experimental): Behavioral Intervention Video
  Interventions: Behavioral: Video

INTERVENTIONS:
Behavioral: Video — Behavioral Intervention Video
  Arms: Video

SUMMARY:
The design of this randomized controlled trial (RCT) is to test the effectiveness of a post-test behavioral video in educating adolescents about HIV transmission and affecting their intentions to engage in risk-reduction behavior.

DETAILED DESCRIPTION:
Adolescents are at risk for HIV because of their engagement in high risk sexual activity. This study seeks to determine effective ways to educate teens about HIV and how to protect themselves by use of multimedia. All eligible participants who agree to enroll in this trial will be randomized into two arms: the behavioral intervention video (intervention group) or meeting with an in-person counselor (control group) as they wait for their rapid HIV results. The goals of the RCT involve establishing the feasibility of using touch-screen technology for teenagers in the ED; establishing the receptivity of teens to HIV rapid testing in the ED; providing data on rates, and obtaining preliminary data on the effectiveness of the video in changing condom efficacy, condom outcome expectancies and condom use intention. Consenting to rapid HIV testing is a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Youth who have had vaginal, anal or oral sex
2. 15-21 years of age
3. English speaking

Exclusion Criteria:

1. Clinically unstable secondary to pain or unstable vitals signs
2. Unable to understand the consent process for the study
3. Known HIV status or recent HIV test
4. Language other than English

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Intention to use condoms | 5 months
  Participants are asked about their intention to use condoms during sexual activity over the next 5 months

SECONDARY OUTCOMES:
Consent to rapid HIV testing | Immediate
  All participants are offered an HIV test but do not have to get tested to participate. We will evaluate whether the videos or counselors convince more participants to get tested for HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Calderon, MD MS, Principal Investigator — Jacobi Medical Center/ Albert Einstein Medical College
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Calderon Y, Cowan E, Leu CS, Brusalis C, Rhee JY, Nickerson J, Leider J, Bauman LJ. A human immunodeficiency virus posttest video to increase condom use among adolescent emergency department patients. J Adolesc Health. 2013 Jul;53(1):79-84. doi: 10.1016/j.jadohealth.2013.01.028. Epub 2013 Apr 9. PMID 23582525